CLINICAL TRIAL: NCT05043064
Title: Validity Evidence for Simulation-based Assessment of Robotic Cardiac Surgical Skills and Examination of Learning Curves in Wet Labs
Brief Title: Robotic Cardiac Surgery Wet Lab Simulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Gennady Atroshchenko, Principal Investigator, Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-000992-55
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Robotic Cardiac Surgery Simulation
Keywords: Robotic Cardiac Surgery; Wet Lab Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All tasks will be recorded and evaluated blinded using the modified Global Evaluative Assessment of Robotic Skills (mGEARS) score by two not participating raters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experienced robotic cardiac surgeons (Active Comparator)
  Interventions: Procedure: Wet lab tasks
- Cardiac surgeons with limited robotic experience (Active Comparator)
  Interventions: Procedure: Wet lab tasks
- Non-cardiac surgeons with limited robotic experience (Active Comparator)
  Interventions: Procedure: Wet lab tasks

INTERVENTIONS:
Procedure: Wet lab tasks — Robotic-assisted internal thoracic artery harvesting, mitral annulus sutures placement and atrial closure in porcine model

SUMMARY:
The goal of this study is to investigate validity of the wet lab robotic cardiac surgery model used for training in robotic cardiac surgery and to evaluate learning curves in trainees of different surgical specialities. The investigators hope to recruit experienced robotic cardiac surgeons (experts) and cardiac and non-cardiac surgeons with minimal robotic experience (trainees). Participants will perform three predetermined tasks common in the wet lab robotic cardiac surgery training. Participants will be evaluated at baseline for each task. From experts' performance the mastery learning level will be calculated. Trainees will perform the tasks until mastery is achieved. The investigators will then be able to evaluate validity of the wet lab model and analyze learning curves in all participants by rating their performance.

ELIGIBILITY:
Inclusion Criteria:

* Experienced robotic cardiac surgeons: robotic surgeons with total volume > 50 robotic cardiac operations and at least 20 robotic cases annually
* Cardiac surgeons with limited robotic experience (robotic novices): on-going or completed cardio-thoracic residency
* Non-cardiac surgeons with limited robotic experience (robotic novices): on-going or completed surgical specialty residency (general surgery, urology, gynaecology, ENT surgery)

Exclusion Criteria:

* Robotic novices with > 5 hours experience of any robotic system

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gennady V Atroshchenko, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Atroshchenko GV, Korup LR, Hashemi N, Ostergaard LR, Tolsgaard MG, Rasmussen S. Artificial intelligence-based action recognition and skill assessment in robotic cardiac surgery simulation: a feasibility study. J Robot Surg. 2025 Jul 13;19(1):384. doi: 10.1007/s11701-025-02563-3. PMID 40652436
- [Derived] Atroshchenko GV, Navarra E, Valdis M, Sandoval E, Hashemi N, Cerny S, Pereda D, Palmen M, Bjerrum F, Bruun NH, Tolsgaard MG. Simulation-based assessment of robotic cardiac surgery skills: An international multicenter, cross-specialty trial. JTCVS Open. 2023 Nov 2;16:619-627. doi: 10.1016/j.xjon.2023.10.029. eCollection 2023 Dec. PMID 38204726

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experienced Robotic Cardiac Surgeons | Cardiac Surgeons With Limited Robotic Experience | Non-cardiac Surgeons With Limited Robotic Experience
Started | 4 | 7 | 8
Completed | 4 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experienced Robotic Cardiac Surgeons | Cardiac Surgeons With Limited Robotic Experience | Non-cardiac Surgeons With Limited Robotic Experience | Total
Number analyzed (Participants) | 4 | 7 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 7 | 17
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [42 to 53] | 55 [43 to 63] | 42 [36 to 48] | 45 [42 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 5
  Male | 4 | 5 | 5 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time-based Score
Description: The time-based score (TBS) was calculated as follows:
  TBS = maximal total training time per task - actual completion time - errors.
  Units of measure - seconds. Minimum score 0, Maximum score 1222.
  TBS was calculated in seconds, where 0 was the lowest score and a higher number indicated a faster time to perform the task.
  The score range
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experienced Robotic Cardiac Surgeons | Cardiac Surgeons With Limited Robotic Experience | Non-cardiac Surgeons With Limited Robotic Experience
Number analyzed (Participants) | 4 | 7 | 8
score on a scale | 553 (47) | 127 (171) | 143 (181)

2. Secondary Outcome: Modified Global Evaluative Assessment of Robotic Skills (mGEARS)
Description: In modified Global Evaluative Assessment of Robotic Skills (mGEARS) the tasks were not rated on autonomy domain as autonomy could not be evaluated from recordings.
  The mGEARS score was used to evaluate the overall robotic proficiency by 5 domains: depth perception, bimanual dexterity, efficiency, force sensitivity, and robotic control. The score ranged from 5 to 25, where 5 and 25 indicated the least and most proficient performance, respectively.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experienced Robotic Cardiac Surgeons | Cardiac Surgeons With Limited Robotic Experience | Non-cardiac Surgeons With Limited Robotic Experience
Number analyzed (Participants) | 4 | 7 | 8
score on a scale | 20 (5) | 13 (2) | 11 (3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Experienced Robotic Cardiac Surgeons | Cardiac Surgeons With Limited Robotic Experience | Non-cardiac Surgeons With Limited Robotic Experience
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT05043064/Prot_SAP_000.pdf